CLINICAL TRIAL: NCT01372592
Title: SpineTRACK (Translating Radiographic and Clinical Knowledge) Registry: Outcomes Data Collection in Degenerative, Deformity, and Trauma Patients
Brief Title: SpineTRACK Registry - Spinal Outcomes Registry
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.REG1101
Record Dates: First submitted 2011-03-25; First posted 2011-06-14 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Vertebra; Degeneration; Spinal Trauma; Spinal Deformity
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Degenerative: Patients being treated for degenerative spine conditions.
  Interventions: Procedure: Surgery
- Deformity: Patients being treated for a deformity spine condition.
  Interventions: Procedure: Surgery
- Trauma: Patients being treated for a trauma related spine condition.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Patients will receive standard of care surgical treatment dependent on his/her spinal condition.

SUMMARY:
The Spine TRACK Spinal Surgery Registry is a prospective multi-center observational data collection initiative, to capture clinical and radiographic outcomes in candidates for spine surgery with degenerative, deformity, and traumatic pathologies. As an observational database, there are no initial driving hypotheses, but rather data will be mined to answer unforeseen questions, but which may include broad topics such as comparative effectiveness between and among various surgical treatment options, and/or outcomes in various subgroups of patients such as defined by demographics, comorbidities, indications and symptoms, treatment variables, and/or outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for spinal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are evaluated and scheduled to undergo surgical treatment for a spine-related condition are eligible to participate in this registry.
Sampling Method: Probability Sample
Enrollment: 8079 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
To create a database of radiographic and clinical outcome measures of spinal surgery patients to evaluate the efficacy of various procedures for multiple diagnoses. | 24 months then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — NuVasive
Locations (28):
- United States (26):
  - Spine Group Arizona, Phoenix, Arizona
  - SD Center for Spinal Disorders, La Jolla, California
  - Orthopaedic Specialty Institute, Orange, California
  - UCSF Dept. of Orthopaedic Surgery, San Francisco, California
  - Durango Orthopaedics, Durango, Colorado
  - University of South Florida Department of Neurosurgery, Tampa General Hospital, Tampa, Florida
  - Piedmont Physicians, Atlanta, Georgia
  - Midwest Orthopaedics at Rush University, Chicago, Illinois
  - OrthoIndy Northwest, Indianapolis, Indiana
  - University of Minnesota Medical, Minneapolis, Minnesota
  - Spine Midwest, Jefferson City, Missouri
  - Spinemore, LLC, St Louis, Missouri
  - Western Regional Center for Brain & Spine Surgery, Surgery Center of S. Nevada, Las Vegas, Nevada
  - Ocean Orthopaedics, Tomas River, New Jersey
  - University of Buffalo, Buffalo, New York
  - Morehead NeuroSpine, Eden, North Carolina
  - Bone & Joint Surgery Clinic, Raleigh, North Carolina
  - Wake Orthopaedics, Raleigh, North Carolina
  - NeuroSpine Institute, Eugene, Oregon
  - Team2 Solutions, LLC, Medford, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Orthopedics & Sports Medicine, Houston, Texas
  - Austin Spine, Lakeway, Texas
  - Salt Lake Orthopedic Clinic, Salt Lake City, Utah
  - NeoSpine, Puyallup, Washington
  - Northwest Orthopaedic Specialists, PS, Spokane, Washington
- Brazil (2):
  - Luis Pimenta, MD, São Paulo, BR
  - Hospital Ortopedico, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.nuvasive.com